CLINICAL TRIAL: NCT02448121
Title: Treatment for Hip, Knee, Ankle and Shoulder Osteonecrosis With Autologous Mononuclear Cells Transplantation in People With Sickle Cell Disease
Brief Title: Autologous Bone Marrow Stem Cell Transplantation for Osteonecrosis in Sickle Cell Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Bahia (Other)
Collaborators: Hospital Universitário Professor Edgard Santos (Other); Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Vitor Fortuna, PhD, Federal University of Bahia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 25000039812/2005-99; 11738 (Registry Identifier: CONEP)
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Avascular Necrosis of Bone; Sickle Cell Disease
Keywords: Cell therapy; Sickle cell disease; Hip Osteonecrosis; Autologous implantation; Mesenchymal stromal cell; Humeral Osteonecrosis; Knee Osteonecrosis; Ankle Osteonecrosis
MeSH Terms: conditions — Osteonecrosis; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous bone marrow stem cell graft (Experimental): Autologous bone marrow stem cell implantation
  Interventions: Procedure: Autologous bone marrow stem cell graft

INTERVENTIONS:
Procedure: Autologous bone marrow stem cell graft — All patients will undergo autologous bone marrow stem cell implantation into the necrotic lesion area using a minimally invasive technique.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of autologous bone marrow stem cells in sickle cell disease patients with osteonecrosis

DETAILED DESCRIPTION:
The aim of this study is to evaluate autologous bone marrow stem cells transplantation as a safe and potentially beneficial treatment for sickle cell disease patients with osteonecrosis.

ELIGIBILITY:
Inclusion Criteria:

* Stable sickle cell disease patients
* FICAT classification of osteonecrosis, inclusive of Stage II.
* Diagnosis will be based on X-Ray and magnetic resonance imaging (MRI).
* No infection in affected bones at the time of surgery.
* Patient competent to give informed consent.
* Scoring at least 20 points on the pain and daily life activities questionnaire.

Exclusion Criteria:

* FICAT stage III or more
* Patients with a history of corticosteroids or on active therapy
* Bone infection at the limb affected by necrosis
* Recurrent painful crises,
* Immunosuppressive drug therapy,
* Pregnancy,
* Presence of neoplastic disease or any other clinical concurrent condition other than sickle cell disease that predisposed them to the development of osteonecrosis of the femoral head

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-08; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in Functional / Clinical Score of 10 points or more | 60 months
  Standardized and objective scoring system to rate patient's functional abilities

SECONDARY OUTCOMES:
Numeric pain intensity scale (0-10) | 60 months
  VAS scoring system
Disease progression defined as progression to a fractural stage of osteonecrosis | 60 months
  Radiographic signals
Reoperation rate | 60 months
  Need for further surgery or hip replacement
Radiological progression | 60 months
  Radiological progression is defined according to the development of the Ficat- and Steinberg-staging system of osteonecrosis. It is based on radiological findings in X-Ray and MRI scans, respectively, and it is useful in predicting outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: GIldasio Daltro, MD, Study Director — Federal University of Bahia; Vitor Fortuna, PhD, Principal Investigator — Federal University of Bahia; Roberto Meyer, MD, Study Chair — Federal University of Bahia; Radovan Borojevic, PhD, Study Chair — Federal University of Bahia

REFERENCES:
- [Background] Hernigou P, Daltro G, Filippini P, Mukasa MM, Manicom O. Percutaneous implantation of autologous bone marrow osteoprogenitor cells as treatment of bone avascular necrosis related to sickle cell disease. Open Orthop J. 2008 Apr 25;2:62-5. doi: 10.2174/1874325000802010062. PMID 19478932
- [Background] Hernigou P, Daltro G, Flouzat-Lachaniette CH, Roussignol X, Poignard A. Septic arthritis in adults with sickle cell disease often is associated with osteomyelitis or osteonecrosis. Clin Orthop Relat Res. 2010 Jun;468(6):1676-81. doi: 10.1007/s11999-009-1149-3. Epub 2009 Nov 3. PMID 19885711
- [Background] Hernigou P, Flouzat-Lachaniette CH, Daltro G, Galacteros F. Talar Osteonecrosis Related to Adult Sickle Cell Disease: Natural Evolution from Early to Late Stages. J Bone Joint Surg Am. 2016 Jul 6;98(13):1113-21. doi: 10.2106/JBJS.15.01074. PMID 27385685
- [Result] Daltro GC, Fortuna V, de Souza ES, Salles MM, Carreira AC, Meyer R, Freire SM, Borojevic R. Efficacy of autologous stem cell-based therapy for osteonecrosis of the femoral head in sickle cell disease: a five-year follow-up study. Stem Cell Res Ther. 2015 May 29;6(1):110. doi: 10.1186/s13287-015-0105-2. PMID 26021713
- [Derived] Daltro G, Franco BA, Faleiro TB, Rosario DAV, Daltro PB, Meyer R, Fortuna V. Use of autologous bone marrow stem cell implantation for osteonecrosis of the knee in sickle cell disease: a preliminary report. BMC Musculoskelet Disord. 2018 May 22;19(1):158. doi: 10.1186/s12891-018-2067-x. PMID 29788942